CLINICAL TRIAL: NCT05116930
Title: Neostigmine and Glycopyrrolate for the Treatment of Post Dural Puncture Headache After Known Dural Puncture With a Tuohy Needle: A Pilot Study
Brief Title: Neostigmine and Glycopyrrolate for the Treatment of Headache After Dural Puncture
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark D. Rollins, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-009530
Record Dates: First submitted 2021-11-02; First posted 2021-11-11 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Neostigmine; Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Postpartum dural puncture headache following dural puncture from Tuohy needle (Experimental): Subjects identified as experienced a post dural puncture headache after a confirmed dural puncture from a Tuohy needle will receive an IV administration of the study medications neostigmine and glycopyrrolate.
  Interventions: Drug: Neostigmine; Drug: Glycopyrrolate

INTERVENTIONS:
Drug: Neostigmine — IV infusion 20 μg/kg over 10 minutes repeated every 8 hours for a maximum of 3 doses
Drug: Glycopyrrolate — IV infusion 4 μg/kg over 10 minutes repeated every 8 hours for a maximum of 3 doses

SUMMARY:
The purpose of this study is to evaluate Neostigmine and Glycopyrrolate to treat post-dural puncture headache (PDPH) to reduce the proportion of postpartum women with a PDPH requiring epidural blood patch (EBP) who developed a PDPH after accidental dural puncture.

DETAILED DESCRIPTION:
Hypothesis: Neostigmine and glycopyrrolate will reduce the proportion of postpartum women with a PDPH requiring EBP who developed a PDPH after accidental dural puncture with a Tuohy needle.

Background: The post dural puncture headache (PDPH) is a well-documented complication of dural puncture. Depending on a number of factors, the overall incidence of PDPH following dural puncture with an epidural Tuohy needle is typically around 50%, but can be as high as 70% for certain populations (1, 2, 3).

The headache is characterized as frontal or occipital in nature, with a typical onset of 6-72 hours after dural puncture. It is normally exacerbated by the upright position and improved by the supine position. Associated symptoms may include photophobia, nausea, vomiting, dizziness, tinnitus, neck stiffness, decreased hearing and visual changes (2). These symptoms tend to be extremely debilitating in affected patients, severely limiting their functional capacity until the resolution of the headache (2). The compromise is even greater in postpartum women who also need to care for a newborn, as the time after birth is important for forming attachment and encompasses many new obligations for the new mother.

The treatment of the PDPH often begins with conservative treatment including supportive therapies such as hydration, bed rest, acetaminophen, NSAIDs, and oral opioids. In addition, some evidence exists for the use of caffeine (1,2). While these do not hasten recovery, they may improve symptoms. For PDPH of all etiologies, 72% will resolve spontaneously in 7 days and 89% by 14 days (1).

For patients with moderate to severe symptoms or long lasting headaches, the gold standard for treatment of headaches that do not resolve is the epidural blood patch (EBP) (1,2,4). This treatment has been shown to be effective in 70-98% of patients (1,2,4). However, it has numerous contraindications including fever, infection, coagulopathy, active neurological disease, patient refusal. In addition, a potential complication is yet another dural puncture. Also, while the EBP is generally very safe, it is an invasive procedure with its own complications; it has been associated with very rare but serious complications including: moderate long-lasting backache, meningitis, epidural abscess formation, epidural hematoma formation, and neurologic deficit development (5-8).

The use of neostigmine and atropine in the treatment of PDPH was first described in a randomized placebo-controlled trial in 2018 (9). The addition of neostigmine and atropine to conservative treatment for PDPH resulted in all 41 patients in the treatment group reporting a visual analog scale (NRS) score ≤ 3 after 2 doses, no recurrence of headache, and none receiving EBP. Seven out of 42 (15.9%) patients in the placebo group reported a persistent NRS ≥ 5 and all received EBP. Postulated mechanisms of action of neostigmine and atropine in the treatment of PDPH include increased CSF volume and cerebral vasoconstriction. Patients enrolled in this study developed a PDPH after spinal anesthesia using a 22-gauge Quincke needle. The effects of neostigmine and atropine on PDPH resulting from accidental dural puncture with a larger-bore, 17-gauge epidural Tuohy needle are unknown (9,10).

Neostigmine and atropine, when given concomitantly, antagonize each other's adverse effects resulting in a favorable safety profile (12,13). The most common adverse effects reported include blurred vision, dry mouth, abdominal cramps, muscle twitches, and urinary urgency - all of which were transient (9,11). Additionally, simultaneous administration of neostigmine and atropine likely have a net neutral effect on oxytocin release and likely do not affect lactation or breastfeeding for the mother (14). Both neostigmine and atropine are excreted in very small amounts in the breastmilk and are unlikely to affect the breastfed infant more than transiently (15-16).

In the available literature, the main driver of this improvement is thought to be from the cholinergic effects of neostigmine (9). When unopposed, these cholinergic effects are known to cause side effects such as muscle cramping. The main purpose of adding of atropine in the original study - as well as the addition of an anticholinergic in most clinical practice applications - to neostigmine is to counteract these potential cholinergic adverse reactions. Glycopyrrolate is the anticholinergic of choice for use with neostigmine as a muscle relaxant reversal agent. This is because glycopyrrolate has a pharmacokinetic profile that mirrors neostigmine and is able to more effectively to eliminate the cholinergic effects in patients who receive neostigmine over the duration of the neostigmine pharmacologic effect (17).

Number of Participants: Enrollment of 36 with goal of 18 evaluable patients

Design: Prospective Pilot Study

Recruitment: In person contact by OB Anesthesia resident, OB Anesthesia fellow, Anesthesia consultant, or Research Coordinator

Recruitment process: Patients will be identified as at risk on the labor and delivery ward after they have experienced a known dural puncture with a Tuohy needle. Patients will be assessed daily while in the hospital for signs and symptoms of a PDPH. If patient meets criteria after dural puncture (a positional headache after known dural puncture, worsened by the upright position, NRS score of ≥ 4), they will be informed of the study procedures, given time to ask questions regarding procedures, and decide if they consent to participation. Patients will also be counseled on the risks and benefits of EBP and can elect to proceed with EBP at any point in the study.

Intervention:

Parturients with a PDPH after documented accidental dural puncture with a Tuohy needle and a NRS score of ≥ 4 will receive a slow infusion of 20 μg/kg neostigmine and 4 μg/kg glycopyrrolate IV given over 10 minutes. Patients will be monitored with blood pressure measurements every 3 minutes along with continuous EKG and pulse oximetry during the infusion and for 20 minutes after completion of the infusion. This regimen is repeated every 8 hours for a maximum of 3 doses. Treatments continue until a NRS score ≤ 3 is achieved or the patient elects to proceed with an epidural blood patch. Patients also receive conservative PDPH management which includes encouraging oral hydration, encouraging oral caffeine consumption in patients who regularly consume caffeine, 1 g acetaminophen every 6 hours, and 600 mg ibuprofen every 6 hours. Oxycodone 5-10 mg every 4 hours PRN may be utilized for postoperative pain.

Safety Monitoring: Patients receiving the intervention will be monitored during and after the intervention for abdominal or muscle cramps, blurred vision, dry mouth, or urinary urgency by the OB anesthesia provider administering the intervention. They will be instructed to call the research PI if they have any of these complications. Patients will also be monitored with blood pressure measurements every 3 minutes along with continuous EKG and pulse oximetry during the infusion and for 20 minutes after completion of the infusion.

Consent process: Consent will be obtained after identification of a PDPH after documented accidental dural puncture with a Tuohy needle and a NRS score of ≥ 4 in the patient's hospital room. Patients will be given sufficient time to ask any questions to the attending/resident anesthesiologist and research personnel related to the procedure and this research study.

ELIGIBILITY:
Inclusion Criteria:

* Post-dural puncture headache (PDPH) after documented dural puncture with Tuohy needle during placement of epidural analgesia for labor and no other explanation for headache (HA).
* Onset of HA within 72 hours of delivery.

Exclusion Criteria:

* Patient refusal.
* Visual analog scale (NRS) score < 4.
* History of migraine headaches.
* Asthma.
* Arrhythmia.
* Heart block.
* Myasthenia gravis.
* Inability to understand pain scores and other questionnaires.
* Inability to speak English.
* Contraindication to acetaminophen or NSAIDs.
* Temperature > 38.5 C.
* Prior EBP done for this HA.

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of postpartum women requiring epidural blood patch | 2 weeks
  Total number of postpartum women with a post dural puncture headache (PDPH) requiring epidural blood patch (EBP)

SECONDARY OUTCOMES:
Change in pain scores | Baseline, 1 hour, 8 hours, 16 hours, 24 hours, 48 hours, 1 week, and 2 weeks after intervention
  Measured using the Numeric Rating Scale (NRS) pain score (0-10) with patient in sitting position for 5 min
Adverse Events | 2 weeks
  Total number of adverse events experienced by subjects

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rollins, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turnbull DK, Shepherd DB. Post-dural puncture headache: pathogenesis, prevention and treatment. Br J Anaesth. 2003 Nov;91(5):718-29. doi: 10.1093/bja/aeg231. PMID 14570796
- [Background] Amorim JA, Gomes de Barros MV, Valenca MM. Post-dural (post-lumbar) puncture headache: risk factors and clinical features. Cephalalgia. 2012 Sep;32(12):916-23. doi: 10.1177/0333102412453951. Epub 2012 Jul 27. PMID 22843225
- [Background] Flaatten H, Rodt S, Rosland J, Vamnes J. Postoperative headache in young patients after spinal anaesthesia. Anaesthesia. 1987 Feb;42(2):202-5. doi: 10.1111/j.1365-2044.1987.tb03001.x. PMID 3826597
- [Background] Abouleish E, Vega S, Blendinger I, Tio TO. Long-term follow-up of epidural blood patch. Anesth Analg. 1975 Jul-Aug;54(4):459-63. doi: 10.1213/00000539-197554040-00012. PMID 125053
- [Background] Cornwall RD, Dolan WM. Radicular back pain following lumbar epidural blood patch. Anesthesiology. 1975 Dec;43(6):692-3. doi: 10.1097/00000542-197512000-00023. No abstract available. PMID 127535
- [Background] Mehta SP, Keogh BP, Lam AM. An epidural blood patch causing acute neurologic dysfunction necessitating a decompressive laminectomy. Reg Anesth Pain Med. 2014 Jan-Feb;39(1):78-80. doi: 10.1097/AAP.0000000000000025. PMID 24310044
- [Background] Reynolds AF Jr, Hameroff SR, Blitt CD, Roberts WL. Spinal subdural epiarachnoid hematoma: a complication of a novel epidural blood patch technique. Anesth Analg. 1980 Sep;59(9):702-3. No abstract available. PMID 7191232
- [Background] Sperry RJ, Gartrell A, Johnson JO. Epidural blood patch can cause acute neurologic deterioration. Anesthesiology. 1995 Jan;82(1):303-5. doi: 10.1097/00000542-199501000-00038. No abstract available. PMID 7832316
- [Background] Abdelaal Ahmed Mahmoud A, Mansour AZ, Yassin HM, Hussein HA, Kamal AM, Elayashy M, Elemady MF, Elkady HW, Mahmoud HE, Cusack B, Hosny H, Abdelhaq M. Addition of Neostigmine and Atropine to Conventional Management of Postdural Puncture Headache: A Randomized Controlled Trial. Anesth Analg. 2018 Dec;127(6):1434-1439. doi: 10.1213/ANE.0000000000003734. PMID 30169405
- [Background] Nair AS. Questions Regarding the Use of Neostigmine-Atropine to Treat Postdural Puncture Headache. Anesth Analg. 2019 Jun;128(6):e126-e127. doi: 10.1213/ANE.0000000000004156. No abstract available. PMID 31094821
- [Background] Daoud M, Asfour M, Mubashirulhassan S. Missed Neostigmine-Atropine Side Effects: Uncommonly Noticed Postanesthesia but Commonly Noticed in Other Situations. Anesth Analg. 2019 Jun;128(6):e128. doi: 10.1213/ANE.0000000000004158. No abstract available. PMID 31094823
- [Background] Abrishami A, Ho J, Wong J, Yin L, Chung F. Sugammadex, a selective reversal medication for preventing postoperative residual neuromuscular blockade. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD007362. doi: 10.1002/14651858.CD007362.pub2. PMID 19821409
- [Background] Chrapkiewicz NB, Beale EG, Granner DK. Induction of the messenger ribonucleic acid coding for phosphoenolpyruvate carboxykinase in H4-II-E cells. Evidence for a nuclear effect of cyclic AMP. J Biol Chem. 1982 Dec 10;257(23):14428-32. PMID 6292224
- [Background] Salem MG, Richardson JC, Meadows GA, Lamplugh G, Lai KM. Comparison between glycopyrrolate and atropine in a mixture with neostigmine for reversal of neuromuscular blockade. Studies in patients following open heart surgery. Br J Anaesth. 1985 Feb;57(2):184-7. doi: 10.1093/bja/57.2.184. PMID 2857570
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials
- See also: Statement on Sugammadex during pregnancy and lactation. Soap.org. — https://www.soap.org/assets/docs/SOAP_Statement_Sugammadex_During_Pregnancy_Lactation_APPROVED.pdf
- See also: Drugs and Lactation Database (LactMed) — https://www.ncbi.nlm.nih.gov/books/NBK501922/
- See also: Statement on Resuming Breastfeeding after Anesthesia. Asahq.org. — https://www.asahq.org/standards-and-practice-parameters/statement-on-resuming-breastfeeding-after-anesthesia